CLINICAL TRIAL: NCT06653868
Title: Grafting of the Peri-implant Bony Defects Around Immediate Implants Using Xenogenic Versus Alloplastic Sticky Grafts: Randomized Controlled Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, bassant mohye, bassant mohye, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: per631
Record Dates: First submitted 2024-10-21; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Bone Loss, Alveolar
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Dental Implants

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- immediate implant placement surgery with filling the gap distance with alloplastic sticky graft (Experimental): immediate implant placement surgery with filling the gap distance with injectable platelet rich fibrin combined with alloplast.
  Interventions: Procedure: dental implant with bone augmentation
- immediate implant placement surgery with filling the gap distance with xenogenic sticky bone (Experimental): immediate implant placement surgery with filling the gap distance with injectable platelet rich fibrin combined with xenograft.
  Interventions: Procedure: dental implant with bone augmentation

INTERVENTIONS:
Procedure: dental implant with bone augmentation — gap distance augmentation with bone graft
  Other Names: gap distance augmentation

SUMMARY:
In patients with a single non restorable tooth, does filling the peri-implant buccal gap with alloplastic sticky grafts result comparable results compared to xenogenic sticky grafts?

DETAILED DESCRIPTION:
The buccal aspect of the dental implant has great importance, especially in the aesthetic zone, because the buccal bone is very thin especially in the anterior maxilla and its resorption can result in recession of the soft tissue. A gap occurs in immediately placed implant due to discrepancy between the dimensions of the extraction socket and the implant. Augmentation of the buccal gap decreases the amount of buccal bone resorption and soft tissue recession . Filling the peri-implant defects has been widely discussed to prevent further bone loss. The use of biologic materials such as platelet rich fibrin can enhance the quality of alloplastic bone grafts to give comparable effect when compared to xenogenic grafts.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with healthy systemic condition (Mazzotti et al., 2023).
2. Age from 20-50 years old
3. Patients must be free of any systemic disease which could influence the surgical procedure.
4. Tooth involved in the esthetic zone.
5. Sufficient hard and soft tissue volume in vertical and buccolingual direction
6. Natural teeth adjacent to the involved tooth will be required to be free from infection.
7. Controlled oral hygiene.
8. Indication for tooth extraction included (Degidi et al., 2012);

   * Endodontic failures
   * Untreatable caries
   * Non- restorable teeth
   * Vertical root fracture
   * Remaining roots

Exclusion Criteria:

- 1.Pregnant females 2.Smokers (Khuller, 2009) 3.Unmotivated and uncooperative patients with poor oral hygiene 4.Patients with habits that may compromise the longevity and affect the result of the study as alcoholism or parafunctional habits.

5.Presence of acute dento-alveolar infection.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-20 (Estimated); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
bone changes | 6 months
  superimposition

SECONDARY OUTCOMES:
pink esthetic score | 6 months
  soft tissue esthetics

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided